CLINICAL TRIAL: NCT04824053
Title: Comparative Analysis of the Effects of UNICLA-A2 Against Conventional Dairy Products Administered Daily in Patients At High-risk Colorectal Cancer Development Who Have Undergone Polypectomy
Brief Title: Effects of UNICLA-A2 Dairy Products on Patients At High-risk of Colorectal Cancer Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Cooperativas Lacteas Unidas (Industry); Hospital Clínico Universitario Lozano Blesa (Other)
Responsible Party: Principal Investigator, Ángel Lanas Arbeloa, Head of Digestive Service (University Clinic Hospital Lozano Blesa) and Principal Investigator, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F19-028.0
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Polyp
Keywords: polyp; inflammation; fecal microbiota
MeSH Terms: conditions — Polyps; Inflammation | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UNICLA-A2 milk and its subproducts (Experimental): Participants (n=17) ingest milk and dairy products made from cows homozygous for beta casein A2 during 3 months. These products are also enriched in insaturated fatty acids and selenium. The daily intake reflects the habitual consumption habits. Recommended amounts are 250 mL of milk, a yogurt and 50 g fresh cheese per day.
  Interventions: Dietary Supplement: Milk from genetically selected homozygous- β-casein-A2 cows fed with forages and a concentrate enriched on linseed and selenized yeast as sources of PUFAs and selenium; Dietary Supplement: Yogurt made from milk of genetically selected homozygous- β-casein-A2 cows fed with forages and a concentrate enriched on linseed and selenized yeast as sources of PUFAs and selenium; Dietary Supplement: Fresh cheese made from milk of genetically selected homozygous- β-casein-A2 cows fed with forages and a concentrate enriched on linseed and selenized yeast as sources of PUFAs and selenium
- Placebo (Placebo Comparator): Participants (n=17) ingest conventional dairy products and milk daily during 3 months. As happens in the UNICLA-A2 arm, the daily intake reflects habitual dairy consumption habits in "real life" conditions, without forcing or inducing greater consumption. Therefore, recommended amounts are 250 mL of milk, a yogurt and 50 g fresh cheese per day.
  Interventions: Dietary Supplement: Conventional milk; Dietary Supplement: Conventional yogurt; Dietary Supplement: Conventional fresh cheese

INTERVENTIONS:
Dietary Supplement: Milk from genetically selected homozygous- β-casein-A2 cows fed with forages and a concentrate enriched on linseed and selenized yeast as sources of PUFAs and selenium — The daily intake should reflect habitual consumption habits in "real life" conditions, without forcing or inducing greater consumption. Therefore, patients will be recommended a daily intake of 250 mL of milk. The intervention duration will be 3 months
  Other Names: UNICLA-A2 milk
  Arms: UNICLA-A2 milk and its subproducts
Dietary Supplement: Conventional milk — The daily intake should reflect habitual consumption habits in "real life" conditions, without forcing or inducing greater consumption. Therefore, patients will be recommended a daily intake of 250 mL of milk. The intervention duration will be 3 months
  Arms: Placebo
Dietary Supplement: Yogurt made from milk of genetically selected homozygous- β-casein-A2 cows fed with forages and a concentrate enriched on linseed and selenized yeast as sources of PUFAs and selenium — The daily intake should reflect habitual consumption habits in "real life" conditions, without forcing or inducing greater consumption. Therefore, patients will be recommended a daily intake of one yogurt. The intervention duration will be 3 months
  Other Names: UNICLA-A2 yogurt
  Arms: UNICLA-A2 milk and its subproducts
Dietary Supplement: Conventional yogurt — The daily intake should reflect habitual consumption habits in "real life" conditions, without forcing or inducing greater consumption. Therefore, patients will be recommended a daily intake of one yogurt. The intervention duration will be 3 months
  Arms: Placebo
Dietary Supplement: Fresh cheese made from milk of genetically selected homozygous- β-casein-A2 cows fed with forages and a concentrate enriched on linseed and selenized yeast as sources of PUFAs and selenium — The daily intake should reflect habitual consumption habits in "real life" conditions, without forcing or inducing greater consumption. Therefore, patients will be recommended a daily intake of 50 g of fresh cheese. The intervention duration will be 3 months
  Other Names: UNICLA-A2 fresh cheese
  Arms: UNICLA-A2 milk and its subproducts
Dietary Supplement: Conventional fresh cheese — The daily intake should reflect habitual consumption habits in "real life" conditions, without forcing or inducing greater consumption. Therefore, patients will be recommended a daily intake of 50 g of fresh cheese. The intervention duration will be 3 months
  Arms: Placebo

SUMMARY:
Dietary intervention with UNICLA-A2 milk products containing beta casein A2 protein, and higher levels of omega-3 fatty acids and selenium may contribute to maintain the intestinal integrity, reduce inflammatory processes, normalize the immune system, protect against oxidative damage and equilibrate the gut microbiota in high-risk colorectal cancer patients who have undergone polypectomy

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most frequent cancers in the world and has a significant impact in terms of mortality and health costs. It is estimated that CRC causes around 900,000 deaths annually, mainly due to diagnoses made in advanced stages. Colorectal adenomas (CRA) are precancerous lesions that develop into colorectal cancer following a well-known process into the adenoma-carcinoma sequence. Prevention programs include screening for CRA and removing precancerous lesions by polypectomy, but the high recurrence rates after polypectomy makes it necessary to research on potential chemopreventive agents that may reduce this risk. Dietary recommendations or chemoprevention with different nutritional substances (diets rich in fiber, or poor in red meat, etc) or pharmacological substances including vitamin D, calcium, fatty acids, salicylic acetyl acid, nonsteroidal anti-inflammatory agents (NSAIDs), etc) have been studied. In this way, it seems reasonable to evaluate the effect caused by the administration of certain nutrients that affect lipid and protein metabolism involved in cellular homeostasis, in the preservation of the colonic mucosa or the development of lesions may have in populations at risk.

UNICLA A2 dairy products have a different nutrient profile than conventional ones. UNICLA A2 products have higher content in unsaturated fats, that is to say, increased content of healthy fatty acids such as oleic, linolenic, eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA) and conjugated linoleic acid (CLA). Previous studies have suggested a contribution of ω-3 polyunsaturated fatty acids (PUFAs) to reduce pro-inflammatory markers and, have shown they have antimicrobial and negative properties in relation to biofilm formation. These types of biofilm structures are characteristic of proximal CRC. For these reason, ω-3 PUFAs it is thought that they could modify the altered intestinal microbiota in patients at high risk of CRC towards a less pathogenic environment, correcting the gut dysbiosis. Moreover, they have higher selenium levels (Se), an element with essential biological functions which has been suggested improving effects in combination with other anticancer agents in CRC and taking part in the modulation of several processes, such as the immune response, apoptotic cell death, DNA repair, response to oxidative stress, carcinogenic metabolism, tumorigenesis and angiogenesis. Finally, they contain type A2 beta casein, which differs from A1 beta casein by a single amino acid at position 67 of a 107 amino acid chain. This fact is very important because beta casein contains a chain of amino acids called "beta casomorphin" (BCM7) with negative health effects reported. The proline 67 in beta casein A2 has a strong bond with BCM7 that does not allow it to separate and flow freely in milk to be absorbed. However, the mild bond due to histidine 67 in beta casein A1 allows BCM7 to reach the intestinal wall and be absorbed, being associated with intestinal discomfort, gastrointestinal transit time and stool consistency disturbances, abdominal pain and, increased levels of some inflammatory markers.

For these reasons, in this proposal the investigators aim to determine whether the change from conventional dairy products to UNICLA-A2 products but maintaining the habitual consumption habits in "real life" conditions, without forcing or inducing greater consumption, will have positive effects on maintaining the intestinal integrity by reducing the inflammatory profile, and leading the gut microbiota to a less pathogenic environment in patients at high-risk of CRC development.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed with high-risk polyps in the colorectal cancer screening programme or in the relative's colon cancer prevention program or patients who are in follow-up due to prior detection of polyps with any of the following characteristics:

   * At least 10 adenomas
   * At least 5 proximal serrated polyps (PSP)
   * At least 2 serrated polyps with diameters ≥10 mm
   * Serrated Polyposis Syndrome (SPS)
   * Early invasive CRC (stage pT1) endoscopically resected (surgery not required)
   * A sessile or flat lesion ≥ 20 mm with fragmented resection
   * Patients with previous resection of polyps in which the resection margin was not assessable and are considered susceptible to repeat colonoscopy
   * Patients with intramucosal carcinoma in situ or invasion of the lamina propria (pTis)
2. Regular consumer of milk and dairy products.
3. Informed consent form signed.

Exclusion Criteria:

1. History of allergic reaction attributed to compounds of similar chemical composition to the study agents.
2. Incomplete colonoscopy or with poor quality criteria, Boston <6.
3. Concomitant acetylsalicylic acid (ASA), NSAIDs, misoprostol, corticosteroids or statins needed on a regular or predictable basis during the time of the study.
4. Previous gastrointestinal surgery (colon or small intestine or gastric) that affects the absorption of nutrients.
5. History of familial adenomatous polyposis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline levels in pro-inflammatory circulating markers C-reactive protein (CRP), interleukin (IL)-6, macrophage inhibitory cytokine 1 (MIC-1) and tumour necrosis factor alpha (TNFα), as well as in fecal calprotectin. | At baseline, at 3 months and through study completion, an average of 1 year after the colonoscopy that motivated the patient´s inclusion
  The C-reactive protein and calprotectin are measured by conventional methods in the University Clinic Hospital Lozano Blesa and the circulating biomarkers IL-6, MIC-1 and TNFα by enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Change from baseline in fecal microbiota. | At baseline, at 3 months and through study completion, an average of 1 year after the colonoscopy that motivated the patient´s inclusion
  Stool samples are collected for DNA extraction and ulterior metagenomic analysis of the fecal microbiota's composition. Library construction is carried out with the Ion 16S™ Metagenomics Kit which permits PCR amplification of hypervariable regions of the 16S rDNA gene from bacteria and the material obtained is subjected to next-generation sequencing (NGS) to see the proportions of the main groups of microorganisms in the sample.
To assess the effect of treatment on colorectal adenoma recurrence | Through study completion, an average of 1 year after the initial colonoscopy that motivated the suitability of patients inclusion.
  The number of participants in each arm who develop one or more colorectal adenomas is determined in the follow-up colonoscopy (adenoma detection rate), as well as the presence of advanced or not advanced adenomas, serrated polyps, subtype, location and the total number of adenomas per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Lanas Arbeloa, MD, PhD, Principal Investigator — University Hospital Lozano Blesa. IIS Aragón. CIBER de Enfermedades Hepáticas y Digestivas.
Locations (1):
- Angel Lanas Arbeloa, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MedlinePlus is a service of the National Library of Medicine (NLM), the world's largest medical library, which is part of the National Institutes of Health (NIH). — https://medlineplus.gov/colorectalcancer.html